CLINICAL TRIAL: NCT01370213
Title: Multi-Center Phase II Trial of NK Cell Based Non-Myeloablative Haploidentical Transplantation for Patients With High-Risk Acute Myeloid Diseases
Brief Title: NK Cell Based Non-Myeloablative Transplantation in Acute Myeloid Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011LS027; MT2011-05 (Other: Blood and Bone Marrow Transplant Program)
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: non-myeloablative haploidentical transplant; hematopoietic cell transplant; natural killer cells; adoptive cellular therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine phosphate; Cyclophosphamide; Radiation; IL32 protein, human; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD34 Schema - High-Risk Acute Myeloid Disease (Experimental): Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and filgrastim mobilized CD34+ selected peripheral blood stem cell graft from the same donor.
  Interventions: Drug: Preparative Regimen; Biological: NK Cells; Drug: Interleukin-2; Biological: CD34 Graft/Anti-thymocyte globulin
- TCRα/β Schema - High-Risk Acute Myeloid Disease (Experimental): Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and same donor TCR α/β-depleted cells infusion.
  Interventions: Drug: Preparative Regimen; Biological: NK Cells; Drug: Interleukin-2; Biological: Donor TCR α/β-depleted Graft/ATG

INTERVENTIONS:
Drug: Preparative Regimen — Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant, 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pretransplant, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pretransplant,
  Other Names: Fludara; Cytoxan; radiation
Biological: NK Cells — CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pretransplant.
  Other Names: Natural Killer cells
Drug: Interleukin-2 — Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion
  Other Names: IL-2
Biological: CD34 Graft/Anti-thymocyte globulin — Single donor filgrastim mobilized CD34+ selected peripheral blood stem cell graft (minimum cell dose of 5 x 10^6/kg) on day 0. Rabbit anti-thymocyte globulin (ATG) will be administered on day -1 (0.5 mg/kg) and day +1 and +2 (2.5 mg/kg) pretransplant per institutional guidelines. ATG dosing not identical for all patients.
  Other Names: ATG
  Arms: CD34 Schema - High-Risk Acute Myeloid Disease
Biological: Donor TCR α/β-depleted Graft/ATG — Single donor TCR α/β-depleted filgrastim-mobilized peripheral blood stem cells (PBSC) graft (minimum cell dose of 5 x 10^6/kg) on day 0. ATG will be administered on days -6 and -5 (3mg/kg) for most patients.
  Other Names: stem cell graft
  Arms: TCRα/β Schema - High-Risk Acute Myeloid Disease

SUMMARY:
This is a phase II multi-institutional therapeutic study of NK-cell based nonmyeloablative haploidentical transplantation for the treatment of high-risk acute myeloid diseases. Enrollment will use a two-stage design. Stage 1 will enroll 15 patients unless an early stopping rule is met. If 9 or more of these first 15 patients achieve leukemia free neutrophil engraftment at day +28 accrual will move to stage 2. In stage 2, an additional 28 patients will be enrolled for a total of 43 patients. Patients will be followed for disease response for 2 years.

DETAILED DESCRIPTION:
A reduced intensity conditioning using Fludara, Cytoxan, and irradiation will start on day -22, followed by infusion of donor NK (natural killer) cells on day-17, 6 doses of interleukin-2 (IL-2) to promote NK expansion (day -17 to day -7), 2 doses of ATG for additional immunosuppression to promote engraftment (day -5 to -4), and infusion of a TCR α/β-depleted same donor graft on day 0.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS)

RAEB-1 or RAEB-2 fitting within one of the following disease groups:

* Primary induction failure (PIF): Patients who have not achieved a complete remission (CR) after two induction cycles of cytotoxic therapy (i.e. 7+ 3, MEC, FLAG, etc.) and having ≤ 10,000 absolute circulating blasts measured at least 21 days from prior therapy. Hydroxyurea may be used to control blasts count. Demethylating agents do not count as induction therapy; however early re-induction therapy based on residual disease on a day 14 BM will count as a 2nd cycle
* Relapsed Disease with low disease burden (AML or MDS with ≤ 10,000 absolute circulating blasts. No re-induction attempts are required, but a maximum of 2 reinduction attempts are allowed to be eligible.
* CR3 or greater: This will include CRp defined as CR without platelet recovery to 100,000/mcL.
* CR1 or CR2 with high risk features: Includes therapy induced, prior MDS or MPD, high risk cytogenetic or molecular phenotype with no available donor (sibling or unrelated adult)

Patients with known prior central nervous system (CNS) involvement are eligible provided that it has been treated and CSF is clear for at least 2 weeks prior to enrollment. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.

* Available related HLA-haploidentical adult donor by at least Class I serologic typing at the A&B locus
* Karnofsky score > 50%
* Adequate organ function within 28 days of study registration defined as:

  * Hepatic: AST ≤ 3 x upper limit of institutional normal, total bilirubin ≤ 2.0 mg/dl
  * Renal: estimated glomerular filtration rate (GFR) ≥ 50 mL/min/1.73m^2
  * Pulmonary: Oxygen saturation ≥ 90% on room air and DLCOcor ≥ 40%
  * Cardiac: Ejection Fraction ≥ 35% and no uncontrolled angina, severe uncontrolled ventricular or arterial arrhythmias, or any evidence of acute ischemia or active conduction system abnormalities (rate controlled atrial fibrillation is not an exclusion)
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to NK cell infusion (except for those prescribed as part of the study)
* Women of child bearing potential must have a negative pregnancy test within 28 days prior to study registration and agree to use adequate birth control during study treatment
* Voluntary written consent

Exclusion Criteria:

* Biphenotypic leukemia
* Allogeneic transplant for AML within previous 6 months
* New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan that has not been evaluated with bronchoscopy, if feasible. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Uncontrolled bacterial, fungal or viral infections including HIV - chronic asymptomatic viral hepatitis is allowed
* Known hypersensitivity to any of the study agents
* Received any investigational drugs within the 14 days before 1st dose of fludarabine
* Requires agents other than hydroxyurea to control blast count

Donor Selection:

* Related donor (sibling, parent, offspring, parent or offspring of an HLA identical sibling) 12-75 years of age. (It is recognized individual institutions may have differing donor age guidelines. This is acceptable as long as no donor is younger than 12 years or older than 75 years).
* Body weight of at least 40 kilograms
* In general good health as determined by the medical provider
* HLA-haploidentical donor/recipient match by at least Class I serologic typing at the A&B locus
* Able and willing to have up to 4 separate apheresis collections
* Not pregnant
* Voluntary written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- CD34+ Selection Schema : High-Risk Acute Myeloid Disease: Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and filgrastim mobilized CD34+ selected peripheral blood stem cell graft from the same donor.
  Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant (pre-tx), 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pre-tx, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pre-tx NK Cells: CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pre-tx Interleukin-2: Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion Anti-thymocyte globulin: rabbit anti-thymocyte globulin will be administered on day -6 (0.5 mg/kg) and day -5 (3 mg/kg/day) pre-tx.
- TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease: Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and TCR α/β-depleted haploidentical graft from the same donor.
  Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant (pre-tx), 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pre-tx, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pre-tx NK Cells: CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pre-tx Interleukin-2: Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion Anti-thymocyte globulin: rabbit anti-thymocyte globulin will be administered on day -6 (0.5 mg/kg) and day -5(3 mg/kg/day) pre-tx.
- TCR α/β Depletion and ATG at Different Time Schema: PPatients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and TCR α/β-depleted haploidentical graft from the same donor.
  Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant (pre-tx), 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pre-tx, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pre-tx NK Cells: CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pre-tx Interleukin-2: Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion Anti-thymocyte globulin: rabbit anti-thymocyte globulin will be administered (3 mg/kg/day) pre-tx on different days per institutional guidelines
Period: Overall Study
Arm/Group | CD34+ Selection Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion and ATG at Different Time Schema
Started | 7 | 17 | 1
Completed | 6 | 15 | 1
Not Completed | 1 | 2 | 0
Not completed — Early Death | 1 | 0 | 0
Not completed — Not evaluable | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- CD34+ Selection Schema : High-Risk Acute Myeloid Disease: Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and filgrastim mobilized CD34+ selected peripheral blood stem cell graft from the same donor.
  Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant (pre-tx), 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pre-tx, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pre-tx NK Cells: CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pre-tx Interleukin-2: Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion Anti-thymocyte globulin: rabbit anti-thymocyte globulin will be administered on day -6 (0.5 mg/kg) and day -5(3 mg/kg/day) pre-tx.
- TCR α/β Depletion and ATG at Different Time Schema: Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and TCR α/β-depleted haploidentical graft from the same donor.
  Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant (pre-tx), 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pre-tx, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pre-tx NK Cells: CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pre-tx Interleukin-2: Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion Anti-thymocyte globulin: rabbit anti-thymocyte globulin will be administered (3 mg/kg/day) pre-tx on different days per institutional guidelines
- Total: Total of all reporting groups
Arm/Group | CD34+ Selection Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion and ATG at Different Time Schema | Total
Number analyzed (Participants) | 7 | 17 | 1 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 0 | 14
  >=65 years | 4 | 6 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 0 | 6
  Male | 6 | 12 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Donor Neutrophil Engraftment
Description: The rate of donor neutrophil engraftment in the absence of leukemia at day +28 will be determined. Successful neutrophil engraftment is defined as an absolute donor-derived neutrophil count of >500 cells/μl. Leukemia free is defined as <5% bone marrow blasts, absence of blasts with Auer rods; absence of extramedullary disease; but cytogenetic or molecular minimal residual disease is allowed.
Time Frame: Day 28
Population: CD34 Schema - out of 7 patients, 2 patients were NA due to leukemia, 1 died, and 1 was not evaluable so 3 were analyzed (4 were not).
  TCRα/β Schema - out of 17 patients, 6 patients were NA due to leukemia, 2 were not evaluable.
  TCRα/β Schema + ATG - 1 patient was given ATG at a different time so their results were reported separately
Measure: Count of Participants; unit: Participants
Groups:
- TCR α/β Depletion and ATG at Different Time Schema: Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and TCR α/β-depleted haploidentical graft from the same donor.
  Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant (pre-tx), 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pre-tx, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pre-tx NK Cells: CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pre-tx Interleukin-2: Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion Anti-thymocyte globulin: rabbit anti-thymocyte globulin will be administered on different days per institutional guidelines
Arm/Group | CD34+ Selection Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion and ATG at Different Time Schema
Number analyzed (Participants) | 3 | 9 | 1
Participants | 3 | 7 | 1

2. Secondary Outcome: Number of Participants With Disease Free Survival
Time Frame: At 6 Months
Population: CD34 Schema - of 7, 1 patient was not evaluable. TCRα/β Schema - of 17, 15 patients evaluable for DFS , 2 patients were not evaluable.
  TCRα/β Schema + ATG at different time - 1 patient given ATG at different time so results reported separately
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Selection Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion and ATG at Different Time Schema
Number analyzed (Participants) | 6 | 15 | 1
Participants | 1 | 6 | 1

3. Secondary Outcome: Number of Participants With Treatment Related Mortality (TRM)
Description: Cumulative incidence will be used to estimate TRM.
Time Frame: At 6 Months
Population: CD34 Schema - of 7 patients, 1 was not evaluable. TCRα/β Schema - of 17 patients, 8 died of disease, 2 did not have TRM at 6 months, 2 were not evaluable.
  TCRα/β Schema + ATG at different time - 1 patient given ATG at different time, results reported separately.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Selection Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion and ATG at Different Time Schema
Number analyzed (Participants) | 6 | 15 | 1
Participants | 2 | 5 | 0

4. Secondary Outcome: Number of Participants Who Relapse
Description: Cumulative incidence will be used to estimate relapse.
Time Frame: 2 Years
Population: CD34 Graft - of 7, 1 patient not evaluable, 2 patients did not clear disease, 2 died before 2 years.
  TCRα/β Schema - of 17, 7 didn't achieve remission, 2 died before 2 years, 2 were not evaluable.
  TCRα/β Schema + ATG at different time - 1 patient received ATG at different time, results reported separately.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34+ Selection Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion and ATG at Different Time Schema
Number analyzed (Participants) | 2 | 6 | 1
Participants | 2 | 6 | 0

5. Secondary Outcome: Number of Participants With Early In Vivo Expansion of Natural Killer (NK) Cells
Description: Successful in vivo donor NK cell expansion will be defined by measuring an absolute circulating donor-derived NK cell count of >100 cells/μl in patient's peripheral blood 12 days after infusion.
Time Frame: Day 12
Population: CD34 Graft - of 7, 1 NA due to missing data/tests not performed, 1 not evaluable.
  TCRα/β Schema - of 17 patients, 15 were evaluable for outcome measure criteria, 2 were not evaluable.
  TCRα/β Schema + ATG at different time - 1 given ATG at different time, results reported separately.
Measure: Count of Participants; unit: Participants
Groups:
- TCR α/β Depletion and ATG at Different Time Schema: Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and same donor TCR α/β-depleted cells infusion.
  Preparative Regimen: Preparative Regimen:
  1) fludarabine 40 mg/m^2 x 4 doses on Days -22 through -19 pretransplant, 2) cyclophosphamide 50 mg/kg x 2 doses on Days -20 and -19 pretransplant, 3) total body irradiation 200 cGy twice a day (BID) (at least 6 hours apart) on Day -18 pretransplant,
  NK Cells: CD3^- CD19^- selected, interleukin-2 (IL-2) activated, haploidentical donor natural killer (NK) cells infused on Day -17 pretransplant.
  Interleukin-2: Interleukin-2 6 million units (MU) subcutaneously (SQ) every other day for 6 doses beginning evening of NK cell infusion
  Anti-thymocyte globulin: rabbit anti-thymocyte globulin will be administered on different days per institutional guidelines
Arm/Group | CD34+ Selection Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion Schema : High-Risk Acute Myeloid Disease | TCR α/β Depletion and ATG at Different Time Schema
Number analyzed (Participants) | 5 | 15 | 1
Participants | 1 | 6 | 1

ADVERSE EVENTS:
Groups:
- High-Risk Acute Myeloid Disease: Patients with high risk acute myeloid disease treated with preparative regimen including Fludara, Cytoxan and total body irradiation followed by haploidentical donor NK cells, Interleukin-2, rabbit anti-thymocyte globulin, and same donor TCR α/β-depleted cells infusion.
  Data is reported in a combined manner because the AE data was originally reported in the older database as a single arm. Data was separated out for the outcome measures because there was still access to this data externally. At this point, we are unable to separate the individual instance of adverse events by arm because we cannot access the source data.
Arm/Group | High-Risk Acute Myeloid Disease
Serious Adverse Events (participants affected / at risk) | 19/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Risk Acute Myeloid Disease (N=25)
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 3
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cytomegalovirus (Infections and infestations) | 3
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Fever (General disorders) | 1
Graft Failure (General disorders) | 1
Heart Failure (Cardiac disorders) | 1
Hypocellular Bone Marrow (General disorders) | 2
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Maculo-Papular Rash (Skin and subcutaneous tissue disorders) | 1
Multi-Organ Failure (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Disease Relapse (General disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Retrobulbar Optic Neuritis (Eye disorders) | 1
Sepsis (Infections and infestations) | 2
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Risk Acute Myeloid Disease (N=25)
Abdominal Pain (Gastrointestinal disorders) | 2
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Creatinine Increased (Investigations) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Eye Irritation (Eye disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 18
Epigastric Pain (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 3
Urinary Frequency (Renal and urinary disorders) | 1
Lethargy (General disorders) | 1
Maculo-Papular Rash (Skin and subcutaneous tissue disorders) | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vivid Dreams (Psychiatric disorders) | 1
Pustular Folliculitis, Scalp (Skin and subcutaneous tissue disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Skin Nodules (Skin and subcutaneous tissue disorders) | 1
Vomiting - Intermittent (Gastrointestinal disorders) | 1
Weight Gain (Investigations) | 3
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Chills (General disorders) | 24
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Edema (General disorders) | 15
Erythema at Central Venous Catheter Site (General disorders) | 1
Eye Infection (Infections and infestations) | 1
Facial, Jaw, Parotid Pain (Musculoskeletal and connective tissue disorders) | 1
Fever (General disorders) | 19
Foot Pain (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 23
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14
Infection, NOS (Infections and infestations) | 1
Infusion Related Reaction (General disorders) | 16
Injection Site Reaction (General disorders) | 13
Leg Weakness (Musculoskeletal and connective tissue disorders) | 1
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 14
Vision Changes, NOS (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No